CLINICAL TRIAL: NCT02630277
Title: Evaluation of Treatment of High riSk proLiferative Diabetic retinopathY With Intravitreal Aflibercept Injection (ELYSIAN)
Brief Title: Evaluation of Treatment of High riSk proLiferative Diabetic retinopathY With Intravitreal Aflibercept injectioN
Acronym: ELYSIAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valley Retina Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELYSIAN
Record Dates: First submitted 2015-12-09; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative Diabetic Retinopathy; High Risk PDR; aflibercept; regression of retinal neovascularization
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): 1:1 Intravitreal Aflibercept Injection once every 4 weeks
  Interventions: Drug: Aflibercept
- Arm 2 (Experimental): Intravitreal of Aflibercept once every 4 weeks for 4 months then as needed (PRN)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal Aflibercept Injection 2.0 mg
  Other Names: Eylea

SUMMARY:
To assess the safety and efficacy of intravitreal aflibercept injection in the regression of retinal neovascularization secondary to high-risk PDR.

To characterize baseline/post-induction/maintenance levels of proinflammatory mediators in patients with high-risk PDR

DETAILED DESCRIPTION:
This study will evaluate two dosing regimens (monthly and PRN following a loading dose) for treatment of PDR with intravitreal aflibercept injection. Additionally, the study will identify biomarker mediators in vitreous fluid present at baseline in patients with PDR and will track over the course of a year their profile changes in response to these two dosing regimens. The treatment regimens will provide information on the biomarker profile with a monthly regimen as well as with a variable regimen. Furthermore, biomarker mediators that may be associated with anti-VEGF responders and non-responders may also be identified. 105 biomarker mediators (cytokines/chemokines) which have been identified as playing a role in PDR in published studies will be profiled in patients with PDR.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible eyes will have active PDR with high risk characteristics (HRC) as defined by the DRS. All eyes must meet at least one or both of the following criteria:

   * Any neovascularization of the disc (NVD) + vitreous hemorrhage
   * Mild neovascularization of the disc (NVD) of at least 1/2 to 1/3 disc area as shown in standard photograph 10A of the DRS
   * Moderate neovascularization of the retina elsewhere (NVE) of at least 1/2 disc area as shown in standard photograph 7 of the DRS + vitreous hemorrhage2. Patient's study eye must be treatment naïve; no history of intravitreal anti-angiogenic treatment, intravitreal steroid treatment, or any laser treatment to study eye
2. 18 years or older males and females with a history of diabetes mellitus and ability to sign informed consent
3. ETDRS visual acuity score greater than or equal to 24 letters (approximately 20/320) and less than or equal to 85 letters (approximately 20/20) by the ETDRS visual acuity protocol at the screening visit
4. Eyes with mild pre-retinal hemorrhage or mild vitreous hemorrhage that does not interfere with clear visualization of the macula and optic disc are eligible for this study

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

1. Presence of moderate or dense PRH or VH that prevents clear visualization of the macula and/or optic disc
2. Presence of either:

   * Significant epiretinal membranes involving the macula, or
   * Proliferative diabetic membranes along the major retinal arcades that are extensive enough to cause either:
   * Significant vitreomacular traction or
   * Significant impairment in visual acuity
   * Presence of any tractional retinal detachment
   * Severe ischemia involving the foveal avascular zone (≥1 disc area) as determined by fluorescein angiography performed at the initial screening visit
   * Significant media opacity (due to cornea, anterior chamber, or lens) precluding clear visualization of the macula or optic disc
   * Presence of neovascular glaucoma with or without hyphema
   * Previous treatment with intravitreal steroid injections in the study eye
   * Previous treatment with topical anti-inflammatory medications in the study eye
   * Previous treatment with peribulbar steroid injections in the study eye
   * Previous PRP/focal laser treatment in the study eye
   * History of vitreoretinal surgery in the study eye
   * Previous treatment with anti-angiogenic drugs in either eye
   * History of idiopathic or autoimmune uveitis in either eye
   * Active ocular inflammation (including trace or above) in the study eye
   * Structural damage to the center of the macula in the study eye that is likely to preclude improvement in VA following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, or organized hard-exudate plaque
   * Ocular disorders in the study eye that may confound interpretation of study results, including retinal vascular occlusion, retinal detachment, macular hole, or CNVM of any cause
   * Concurrent disease in the study eye that would compromise VA or require medical or surgical intervention during the study period
   * Cataract surgery in the study eye, yttrium-aluminum-garnet (YAG) laser capsulotomy, or any other intraocular surgery
   * Aphakia or absence of the posterior capsule in the study
   * Uncontrolled glaucoma or previous filtration surgery in the study eye
   * Evidence at examination of infectious blepharitis, keratitis, scleritis or conjunctivitis in either eye or current treatment for serious systemic infection
   * History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 1
   * Participation in an investigational trial within 30 days prior to screening that involved treatment with any drug (excluding vitamins and minerals) or device
   * Pregnancy (positive pregnancy test) or lactation Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Assess ocular and non-ocular adverse events | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Victor H Gonzalez, MD, Principal Investigator — Medical Director